CLINICAL TRIAL: NCT02759042
Title: An Expanded Compassionate Access Protocol for a Single Subject Who Has Completed 24-Weeks of Treatment in PRO140_CD02 Study
Brief Title: An Expanded Access Protocol for a Single Subject Who Has Completed 24-Weeks of Treatment in PR0140_CD02 Study
Acronym: CD02_EA
Status: No longer available | Type: Expanded Access
Sponsor: CytoDyn, Inc. (Industry)
Collaborators: Amarex Clinical Research (Other)
Responsible Party: Sponsor
Other Study IDs: PRO140 CD02_EA
Record Dates: First submitted 2016-04-19; First posted 2016-05-03 (Estimated); Last update posted 2018-03-13 (Actual); Status verified 2017-08

CONDITIONS: HIV
MeSH Terms: interventions — leronlimab

INTERVENTIONS:
Drug: PRO 140 — PRO 140 is a humanized IgG4,κ monoclonal antibody (mAb) to the chemokine receptor CCR5.
  Other Names: PRO140; CCR5 antagonist; Humanized monoclonal antibody to CCR5

SUMMARY:
The primary objective is to provide continued access to PRO 140 to a subject who has completed participation in PRO140_CD02.

DETAILED DESCRIPTION:
This is an open label, single center study designed to provide continued access to PRO 140 to a subject who have completed participation in PRO140_CD02 and continue to receive clinical benefit.

The subject will receive weekly PRO 140 SC injection along with oral ART regimen during the Treatment Phase. The study treatment (PRO 140 SC injections) will be administered by a qualified medical professional or self-administered by the subject.

ELIGIBILITY:
This study will recruit one treatment-experienced, HIV-1 infected patient with CCR5-tropic virus, who has participated in PRO 140_CD02 clinical trial and is continuing to derive clinical benefit from PRO 140 treatment.

Ages: 55 Years to 56 Years | Sex: Male
Age Groups: Adult

CONTACTS AND LOCATIONS:
Overall Officials: Edwin DeJesus, MD, FIDSA, Principal Investigator — Orlando Immunology Center
Locations (1):
- CD02 EA Investigational site, Orlando, Florida, United States